CLINICAL TRIAL: NCT07083505
Title: A Multicenter, Randomized, Open-Label Phase II Clinical Trial Comparing Efficacy and Safety of HB1801 With Taxotere® in Advanced Breast Cancer
Brief Title: A Study Comparing the Efficacy and Safety of HB1801 With Taxotere® in Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-015
Record Dates: First submitted 2025-07-15; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HB1801 (Experimental): HB1801 [administered according to the clinical trial protocol]
  Interventions: Drug: HB1801
- Taxotere® (Active Comparator): Taxotere® 75 mg/ m^2 [administered according to the clinical trial protocol]
  Interventions: Drug: Taxotere®

INTERVENTIONS:
Drug: HB1801 — HB1801 [administered according to the clinical trial protocol]
  Arms: HB1801
Drug: Taxotere® — Taxotere® 75 mg/ m^2 [administered according to the clinical trial protocol]]
  Arms: Taxotere®

SUMMARY:
This is a randomized, open-label, multicenter Phase II clinical trial evaluating the efficacy and safety of HB1801 compared with Taxotere® in patients with advanced breast cancer. A total of 60 subjects with advanced breast cancer are planned to be enrolled.The trial consists of three phases: screening period, open-label treatment period, and follow-up period. HB1801 is Docetaxel for injection (Albumin-bound).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old (based on the date of signing the informed consent form).
* 2. Voluntarily participate in this clinical trial, sign the informed consent form, and be willing and able to adhere to the treatment, visits, and related procedures specified in the protocol.
* 3. Patients with histologically or cytologically confirmed unresectable locally advanced or metastatic breast cancer, meeting the following criteria: a) The investigator determines that the patient is suitable for single-agent docetaxel treatment, in accordance with the 2025 Chinese Society of Clinical Oncology (CSCO) Breast Cancer Treatment Guidelines. b) At least one measurable lesion according to RECIST 1.1 criteria. For lesions previously treated with radiotherapy, the lesion can only be included as a measurable lesion if clear disease progression occurs after radiotherapy.
* 4. Within 7 days before randomization, major organ/system functions are basically normal, meeting the criteria as assessed by laboratory tests.
* 5. ECOG performance status of 0-1 within 7 days before randomization.
* 6. Expected survival time ≥ 3 months.
* 7. For women of childbearing potential (WOCBP): Negative serum pregnancy test within 7 days before randomization. The subject and spouse must agree to use effective contraception from the date of signing the informed consent until 6 months after the last study drug administration. During this period: Female subjects must not be lactating; Male subjects must avoid sperm donation.

Exclusion Criteria:

* 1. Prior treatment with docetaxel monotherapy or combination therapy for unresectable locally advanced or metastatic breast cancer.
* 2. Subjects with partially or completely intestinal obstruction that cannot be relieved by active treatment; history of inflammatory bowel disease, chronic diarrhea, or gastrointestinal bleeding.
* 3. Known severe allergic history or hypersensitivity (NCI-CTCAE v5.0, ≥ grade 3) to human albumin or docetaxel, and/or contraindications; known severe allergic history and/or contraindications to glucocorticoids (including but not limited to active peptic ulcer, severe hypertension, severe hypokalemia, glaucoma, etc.).
* 4. Untreated active brain metastases (including symptomatic brain metastases or leptomeningeal metastases); subjects with treated brain metastases are eligible if the metastatic lesions are stable (brain imaging demonstrates stability for at least 4 weeks before randomization, no new neurological symptoms or neurological symptoms have returned to baseline, and no hormonal therapy is required for at least 14 days before randomization for investigational treatment), and there is no evidence of new or enlarged pre-existing brain metastases.
* 5. History of other malignant tumors within 5 years before randomization, except for cured basal cell carcinoma, squamous cell carcinoma of the skin, or in-situ carcinoma (e.g., cervical in-situ carcinoma).
* 6. Uncontrolled serous effusions (e.g., pleural effusion, ascites, pericardial effusion) requiring frequent drainage or medical intervention within 14 days before randomization, or requiring additional intervention within 2 weeks after intervention (excluding exfoliative cytology of exudates).
* 7. Severe neurological diseases (e.g., epilepsy, dementia) and ≥ grade 3 peripheral neuropathy.
* 8. Severe respiratory diseases, such as asthma requiring glucocorticoid use, chronic obstructive pulmonary disease (acute exacerbation phase), etc.
* 9. History of severe cardiovascular diseases within 6 months before randomization, including but not limited to: 1)Uncontrolled hypertension (defined as sustained systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg despite antihypertensive medication); 2)Severe arrhythmias and conduction abnormalities requiring anti-arrhythmic drugs other than β-blockers or digoxin (except atrial fibrillation and paroxysmal supraventricular tachycardia); 3)History of myocardial infarction, unstable angina, angioplasty, coronary artery bypass surgery; 4)New York Heart Association (NYHA) class II or higher heart failure; 5)QTcF > 480 ms [QTcF = QT/(RR 0.33), where RR is normalized heart rate (60/heart rate)], calculated by Fridericia formula (if abnormal, average three consecutive measurements taken 2 minutes apart); 6)Other clinically significant cardiac diseases as determined by the investigator.
* 10. Severe chronic or active infection requiring intravenous antibacterial, antifungal, or antiviral therapy within 2 weeks before randomization.
* 11. Major organ surgery (except biopsy or infusion device implantation) within 4 weeks before randomization, or scheduled for major organ surgery during the trial.
* 12. Chemotherapy, targeted therapy, immunotherapy, endocrine therapy, or other investigational drugs within 4 weeks or 5 half-lives (whichever is shorter, but at least 2 weeks) before randomization; radiotherapy within 2 weeks before randomization; traditional Chinese medicine with anti-tumor indications within 2 weeks before randomization.
* 13. Unresolved toxicities from prior anticancer therapy to grade 1 or lower (per CTCAE v5.0), except for grade 2 neuropathy, alopecia, hypothyroidism (with hormone replacement), and toxicities determined by the investigator to pose no safety risk.
* 14. Use of strong CYP3A4 inhibitors or inducers within 2 weeks before randomization.
* 15. Vaccination (including live and attenuated live vaccines) within 4 weeks before randomization or planned during the trial.
* 16. Active hepatitis B infection (HBsAg-positive and HBV-DNA > ULN); hepatitis C infection (antibody-positive and HCV-RNA PCR-positive); human immunodeficiency virus (HIV) carrier; active tuberculosis or syphilis infection.
* 17. Concurrent participation in another interventional clinical study, unless participating in an observational (non-interventional) study or follow-up of an interventional study.
* 18. Other conditions deemed by the investigator as unsuitable for trial participation, including but not limited to severe or uncontrolled medical conditions interfering with trial result interpretation or trial compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-10-11 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progressive-free Survival ( PFS) | Up to 18months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 18months
Disease Control Rate (DCR) | Up to 18months
Duration of Response (DoR) | Up to 18months
Overall Survival (OS) | Up to 18months
Incidence and severity of Adverse Events (AEs) | Up to 18months